CLINICAL TRIAL: NCT03178812
Title: The Role of the Cystic Fluid Interleukins 1,8, & 10 and Tumor Necrosis Factor (TNF) Levels in Characterizing Pancreatic Cysts Detected by Endoscopic Ultrasound (EUS)
Brief Title: Role of the Cystic Fluid Interleukins and Tumor Necrosis Factor (TNF) Levels in Characterizing Pancreatic Cysts Detected by Endoscopic Ultrasound (EUS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HYMC-0018-17
Record Dates: First submitted 2017-05-10; First posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: One arm containing patients with pancreatic lesion and one control group arm of healthy volunteers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with pancreatic cysts (Active Comparator): Fine-needle aspiration (FNA) by Endoscopic Ultrasound (EUS) will collect liquid from patients' pancreatic cysts to measure their Interleukin and TNF levels
  Interventions: Procedure: EUS with fine-needle aspiration of pancreatic cyst
- Healthy volunteers (Active Comparator): Laboratory blood test to measure Interleukin and TNF levels
  Interventions: Procedure: EUS with fine-needle aspiration of pancreatic cyst; Diagnostic Test: Laboratory Blood test

INTERVENTIONS:
Procedure: EUS with fine-needle aspiration of pancreatic cyst — EUS with fine-needle aspiration
Diagnostic Test: Laboratory Blood test — Laboratory Blood Test
  Arms: Healthy volunteers

SUMMARY:
This study aims to find a correlation between cytokines levels and malignancy potential of different cystic types.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pancreatic cyst

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Prediction of malignant potential of pancreatic cyst by measuring Interleukin levels | Two years
  Interleukin 1,8,10 will be measured quantitatively by an enzyme-linked immunosorbent assay. The same interleukins levels will be measured in serum of same patients and control group. Results will enable classification of cysts to either high or low risk malignancy potential.
Prediction of malignant potential of pancreatic cyst by measuring TNF levels | Two years
  TNF levels will be measured quantitatively by an enzyme-linked immunosorbent assay. The same TNF levels will be measured in serum of same patients and control group. Results will enable classification of cysts to either high or low risk malignancy potential.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No